CLINICAL TRIAL: NCT01684020
Title: A Prospective, Double-Blinded, Randomized Study Evaluating the Efficacy and Safety of ARTISS Human Fibrin Sealant as Used in External Rhinoplasty
Brief Title: A Study Evaluating the Efficacy and Safety of ARTISS Human Fibrin Sealant as Used in External Rhinoplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DeNova Research (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Steven H. Dayan, Medical Director, DeNova Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ART-RHI-12
Record Dates: First submitted 2012-09-07; First posted 2012-09-12 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Subjects Requesting and Requiring an Open Rhinoplasty
Keywords: rhinoplasty; external rhinoplasty; open rhinoplasty; nose job

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARTISS Human Fibrin Sealant (Experimental): Prior to fixation of the external rhinoplasty skin flap, a thin layer of ARTISS human fibrin sealant will be applied over the nasal tissue and fixated to the skin flap for at least 3 minutes.
  Interventions: Biological: ARTISS human fibrin sealant
- Standard of Care (No Intervention): Fixation of the skin flap created during external rhinoplasty will use the standard of care

INTERVENTIONS:
Biological: ARTISS human fibrin sealant
  Arms: ARTISS Human Fibrin Sealant

SUMMARY:
Rhinoplasty (nasal reconstruction i.e. "a nose job") is a surgical procedure performed on the nose to correct a medical problem or change the appearance of the nose. During the healing process, swelling and/or bruising is likely to occur. A drug called ARTISS Fibrin Sealant may or may not lessen these effects. This study is looking to see the effects of ARTISS on adhering tissue and improving wound healing in an external rhinoplasty. The purpose of this study is to evaluate the safety and effectiveness of rhinoplasty using ARTISS compared to rhinoplasty without using ARTISS in patients undergoing rhinoplasty performed through an external approach.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 65 years of age.
2. Subjects requesting primary rhinoplasty and requiring an external approach.
3. Subjects willing to undergo treatment with fibrin sealant.
4. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
5. Willingness and ability to comply with the PI's standard preoperative and postoperative rhinoplasty instructions.
6. Subjects of childbearing potential must have a negative urine pregnancy test result at Visit 1 and be willing able to use an acceptable method of birth control (e.g., barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following is documented on the medical history:

   * postmenopausal for at least 12 months prior to study drug administration
   * without a uterus and/or both ovaries
   * has had a bilateral tubal ligation for at least 6 months prior to study drug administration.
   * absence of an other physical condition according to the PI's discretion
7. Willingness and ability to provide written photo consent and adherence to photography procedures (i.e., removal of jewelry and makeup).
8. Willingness and ability to provide written informed consent prior to performance of any study related procedure.

Exclusion Criteria:

1. Subjects who are pregnant, nursing, planning to become pregnant, and/or not using a reliable form of birth control.
2. Subjects who are planning a concurrent facial surgery during the operation (eg forehead plasty, blepharoplasty, rhinoplasty, buccal fat removal, any filler injections including fat injections, lip augmentation, skin resurfacing procedures etc.).
3. Subjects with a previous history of rhinoplasty.
4. Subjects with a current history of smoking.
5. Subjects with a previous history of a bleeding or coagulation disorder .
6. Subject with a previous history of a vascular disorder, cardiovascular disease, and/or uncontrolled hypertension.
7. Subjects a previous history of diabetes mellitus with glycosylated hemoglobin (HbA1c) > 7.
8. Subjects undergoing active treatment for a malignancy.
9. Subjects with a previous history of has a connective tissue disorder.
10. Subjects with active or chronic skin disorder.
11. Subjects with a previous history of Bell's palsy.
12. Subjects with a previous history of pathologically or pharmacologically induced immune deficiency.
13. Subjects who have received chronic treatment with immunosuppressive drugs, systemic corticosteroids, or other chronic treatments within 30 days prior to the surgery.
14. Subjects with a known sensitivity to components of FS VH S/D 4 s-apr.
15. Subjects with a previous history of healing complications following previous surgeries (eg, hypertrophic scarring).
16. Subjects with a significant systemic illness or illness localized to the areas of treatment.
17. Subjects with previous history of nasal implants.
18. Subjects with previous or current history of nasal infections.
19. Subjects who have history of blood thinners (aspirin, ibuprofen, naprosyn, herbal supplements, Vitamin E) within the two weeks prior to surgery.
20. Subjects who have smoked within the two weeks prior to surgery.
21. Subjects who have had alcohol or illicit drugs one week prior to surgery.
22. Subjects who have eaten or drank anything after midnight the night prior to surgery.
23. Subjects with current history of chronic drug or alcohol abuse.
24. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
25. Subjects who anticipate the need for surgery, other than the study procedure, or overnight hospitalization during the study.
26. Subjects who, in the Investigator's opinion, have a history of poor cooperation, non compliance with medical treatment or unreliability.
27. Subject has participated in another clinical study involving an investigational product/device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an investigational product/device during the course of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2016-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD, Principal Investigator — DeNova Research
Locations (1):
- DeNova Research, Chicago, Illinois, United States

REFERENCES:
- See also: Related Info — http://www.denovaresearch.com

RESULTS

PARTICIPANT FLOW:
Groups:
- ARTISS Human Fibrin Sealant: Prior to fixation of the external rhinoplasty skin flap, a thin layer of ARTISS human fibrin sealant will be applied over the nasal tissue and fixated to the skin flap for at least 3 minutes.
  ARTISS human fibrin sealant
Period: Overall Study
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 45.3 [18 to 50] | 45.3 [18 to 50] | 45.3 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Edema Severity
Description: Measured at Day 1, 7, 30, 180
  0 None- No apparent edema
  1. Mild- Minimal tissue swelling
  2. Moderate- Moderate edema, nasal features still discernible
  3. Severe- Marked swelling, difficulty distinguishing nasal features
  Scores closer to 0 indicate more favorable results
Time Frame: Measured at Day 1, 7, 30, 180
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
Number analyzed (Participants) | 5 | 5
units on a scale
  Day 1 | 1.25 (1.5) | 1.5 (1.291)
  Day 7 | 1.25 (1.5) | 1 (1.155)
  Day 30 | 1 (0.816) | 1 (1.414)
  Day 180 | 1.25 (1.5) | 0.5 (0.577)

2. Primary Outcome: Median Number of Adverse Events
Description: Safety will be assessed by the incidence of AEs throughout the study period as documented by clinician observations at study visits and in a 30-day subject diary.
Time Frame: 1 day, 1 week, 4 weeks and 6 months following surgery
Measure: Mean (Full Range); unit: number of AE's
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
Number analyzed (Participants) | 5 | 4
number of AE's | 4 [2 to 6] | 10 [8 to 15]

3. Secondary Outcome: Blinded-assessment of Satisfaction
Description: A non-treating blinded evaluator will assess satisfaction with a four-point categorical satisfaction scale [unsatisfied (4), satisfied (3), very satisfied (2), highly satisfied (1))] of subject's grafts using photographs from baseline, 1 month, 3 months, 6 months, and 12 months and will consist of a blinded evaluation in which the physician is aware of the type of graft, but unaware of plating status or the specific grafting site.
  Scores closer to 1 indicate a more favorable outcome
Time Frame: Measured at Baseline, 1 month, 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
Number analyzed (Participants) | 5 | 4
units on a scale
  Baseline | 4 (0) | 4 (0)
  Month 1 | 2.4 (0.894) | 2 (0.816)
  Month 3 | 2 (0) | 1 (0)
  Month 6 | 1.6 (0.894) | 1.33 (0.577)
  Month 12 | 2.5 (0.707) | 2 (0)

4. Secondary Outcome: Objective Ecchymosis Evaluation - PI
Description: The surface area and color of ecchymosis will be evaluated at 1 day, 1 week, 4 weeks, and 6 months following surgery.
  Rating Extent Color 0 No ecchymosis No color change
  1. Up to medial one-third of the lower and/or up eyelid Yellowish color change
  2. Medial half of the upper and/or lower eyelid Light purple
  3. Entire upper and/or lower eyelid Dark purple
  4. Entire part of the lower and upper eyelid and/or conjunctiva Very dark purple
  5. Extension of ecchymosis below the malar bone
  Scores closer to 0 indicate a more favorable outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
Number analyzed (Participants) | 5 | 4
units on a scale
  Day 1 | 1 (1) | 1.5 (0.577)
  Week 1 | 1.4 (0.548) | 0.75 (0.957)
  Week 4 | 0 (0) | 0 (0)
  Month 6 | 0 (0) | 0 (0)

5. Secondary Outcome: Subjective Ecchymosis Evaluation - Subject
Description: Ecchymosis will be determined by a live assessment at 1 day, 1 week, 4 weeks and 6 months following surgery using a six-point categorical edema scale.
  Rating Extent Color 0 No ecchymosis No color change
  1. Up to medial one-third of the lower and/or up eyelid Yellowish color change
  2. Medial half of the upper and/or lower eyelid Light purple
  3. Entire upper and/or lower eyelid Dark purple
  4. Entire part of the lower and upper eyelid and/or conjunctiva Very dark purple
  5. Extension of ecchymosis below the malar bone
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
Number analyzed (Participants) | 5 | 4
units on a scale
  Day 1 | 1 (1) | 2 (0.778)
  Week 1 | 1.5 (0.667) | 2 (0.816)
  Week 4 | 0 (0) | 0 (0)
  Month 6 | 0 (0) | 0 (0)

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Subjects will complete a 30-day diary documenting adverse events such as erythema, pain, tenderness, firmness, swelling, lumps/bumps, bruising, itching and numbness.
Time Frame: Day 30
Measure: Number; unit: participants
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
Number analyzed (Participants) | 5 | 4
participants | 1 | 1

7. Secondary Outcome: Subject Downtime Questionnaire
Description: Subject downtime will be determined using a questionnaire at 1 day, 1 week, 4 weeks, and 6 months following surgery.
  Responders are defined as those subjects experiencing little to no downtime.
  Downtime scale:
  (3) Very Much (2) A Lot
  (1) A Little (0) Not at all
  Scores closer to 0 indicate more favorable outcome
Time Frame: 1 day, 1 week, 4 weeks and 6 months following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
Number analyzed (Participants) | 5 | 4
units on a scale
  Day 1 | 3.4 (0.864) | 4 (0)
  Week 1 | 3.2 (0.447) | 3.25 (0.5)
  Week 4 | 2.4 (1.14) | 2 (0.816)
  Month 6 | 1.2 (0.447) | 1 (0)

8. Secondary Outcome: HPSS Assessment
Description: Changes in subject self-esteem will be determined by subject completion of the Heatherton & Polivy State Self-Esteem (HPSS) Scale at 1 week, 4 weeks and 6 months following surgery.
  HPSS: scored between 1-5 for 20 questions with a total possible score between 20-100
  1. - Not at all
  2. - A little bit
  3. - Somewhat
  4. - Very much
  5. - Extremely
  Scores closer to 100 indicate a more favorable outcome
Time Frame: 1 week, 4 weeks and 6 months following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
Number analyzed (Participants) | 5 | 4
units on a scale
  Week 1 | 3.2 (0.447) | 3.25 (0.5)
  Week 4 | 2.4 (1.14) | 2 (0.816)
  Month 6 | 1.2 (0.447) | 1 (0)

9. Secondary Outcome: Ease of Use
Description: Ease of use will be determined by the treating investigator using a 10 cm Visual Analog Scale (VAS) to demonstrate technical ease.
  (10) - Very diffiucult - (100) - Very easy
  Scores closer to 100 indicate a more favorable outcome
Time Frame: Immediately Post Surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
Number analyzed (Participants) | 5 | 4
units on a scale | 17.6 (5.225) | 39 (17.682)

ADVERSE EVENTS:
Arm/Group | ARTISS Human Fibrin Sealant | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 1/5 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARTISS Human Fibrin Sealant (N=5) | Standard of Care (N=4)
Ecchymosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — A discoloration of the skin resulting from bleeding underneath, typically caused by bruising

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No